CLINICAL TRIAL: NCT05916118
Title: A Phase I, Pilot Study, Single-group Investigating the Feasibility of Exercise During Oxaliplatin Infusions.
Brief Title: Exercise and Oxaliplatin-induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Natasha Dhawan, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY02001529
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise and Oxaliplatin-induced peripheral neuropathy (Experimental): A single arm to evaluate the feasibility and acceptability of having patients exercise during oxaliplatin infusions in the infusion center. Arm will enroll patients receiving oxaliplatin-containing chemotherapy for gastrointestinal cancer or for cancer of unknown primary.
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Patients will be asked to engage in aerobic exercise using a pedal machine to move their arms and legs while in a seated position. Patients will be asked to exercise for a total of 30 minutes, which may be divided in up to three, ten-minute bouts of exercise.

SUMMARY:
This single group study was conducted to test the feasibility and acceptability of implementing an exercise intervention during oxaliplatin infusion across three months of oxalipatin-based chemotherapy in patients with gastrointestinal malignancies.10 patients were enrolled onto this study and validated questionnaires were used to evaluate the feasibility and acceptability of the intervention and collect patient-reported outcomes over the course of study enrollment.

DETAILED DESCRIPTION:
The proposed study is a single arm study to evaluate the feasibility and acceptability of having patients exercise while receiving oxaliplatin infusions in the infusion center. The study will enroll patients receiving oxaliplatin-containing chemotherapy for gastrointestinal cancersor for cancer of unknown primary.

Patients will be provided with a wrist heart rate monitors to be used during the infusions. They will wear the heart monitors during the entirety of the oxaliplatin chemotherapy infusion. Patients will be asked to engage in aerobic exercise using a pedal machine to move their arms and legs while in a seated position. Patients will be asked to exercise for a total of 30 minutes, which will be divided into three, ten minute bouts of exercise, spaced out in 30 minute blocks of time.

The comprehensive surveys including EORTC-QLC-CIPN20 and PROMIS-29 QOL will be completed at baseline, ~6-8 weeks into treatment, and at ~12-14 weeks after treatment initiation. The feasibility and acceptability instruments will be administered ~6-8 weeks into treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving care at Dartmouth-Hitchcock Medical Center in Lebanon, NH
2. Age >18 years
3. Eastern Cooperative Oncology Group Status 0 to 2;
4. Diagnosed gastrointestinal cancer of any stage
5. Scheduled to receive at least 4 cycles of oxaliplatin
6. Complete the International Physical Activity Questionnaire score equal to or greater than 99 MET minutes/week (equivalent to ~30 minutes of walking)
7. Have mediport access prior to enrollment in the study

Exclusion Criteria:

1. Exercise- or mobility-limiting cardiovascular, pulmonary, musculoskeletal, or psychological disease, based on the EMR (electronic medical record) past medical history and/or based on consultation with the medical oncologist;
2. Scheduled major surgery during the study time period;
3. Pre-existing peripheral neuropathy prior to chemotherapy;
4. Patient with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
5. Prior history of treatment with oxaliplatin, docetaxel, or paclitaxel
6. Pregnant women;
7. Prisoners;
8. Inability to read or speak English/unable to consent;
9. Prognosis of less than six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluating the feasibility (adherence) of the intervention by patients | 14 weeks
  * 70% of patients completing >60% of the exercise sessions during all infusion session
  * 60% of patients identifying "agree" or "strongly agree" on the Feasibility of Intervention Measure (FIM), a validated instrument
Evaluating the acceptability of the intervention by patients | 14 weeks
  ≥60% of patients identifying "agree" or "strongly agree" on the Acceptability of Intervention Measure (AIM), a validated instrument

SECONDARY OUTCOMES:
Observe trends of exercise via questionnaires at various time points | 14 weeks
  Observe trends of exercise on patient-reported chemotherapy-induced peripheral neuropathy (via EORTC-QLQ-CIPN20) over time: at baseline, ~6-8 weeks from treatment initiation, and ~12-14 weeks from treatment initiation
Describe changes in quality of life via questionnaires | 14 weeks
  Describe changes in quality of life (via PROMIS-29 QOL) over time: at baseline, ~6-8 weeks from treatment initiation, and ~12-14 weeks from treatment initiation.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth Health, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: Undecided